CLINICAL TRIAL: NCT03869203
Title: Prospective Randomized Controlled Trial of Impact of Enhanced Recovery After Surgery(ERAS) for Outcomes of Total Knee and Hip Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2019-0010
Record Dates: First submitted 2019-03-06; First posted 2019-03-11 (Actual); Last update posted 2019-05-13 (Actual); Status verified 2019-05

CONDITIONS: Arthroplasty, Replacement, Knee, Hip
MeSH Terms: interventions — Enhanced Recovery After Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced recovery after surgery (ERAS) patients (Experimental): Patients planned to undergoing total knee arthroplasty or total hip arthroplasty, following the ERAS perioperative care.
  Interventions: Other: Enhanced recovery after surgery (ERAS)
- Control patients (No Intervention): Patients planned to undergoing total knee arthroplasty or total hip arthroplasty, following the traditional perioperative care.

INTERVENTIONS:
Other: Enhanced recovery after surgery (ERAS) — The patients in the ERAS group were given a pre-treatment drug [300 mg (gabapentin, Neurontin 300mg) and 10 mg oxycontin (oxycontin, Oxycontin CR 10mg) and 2 mg prednisolone (prednisolone 10 mg, Solondo 5mg)] on the evening before surgery. And pre-operative fasting should not exceed 6 hours, and clear liquid fasting should not exceed 2 hours. In addition, 400 ml of oral carbohydrate should be taken 2 to 4 hours before surgery to ensure adequate blood sugar and encourage regular diet (light meal) as soon as possible within a tolerable range after surgery. The initial pain after surgery is actively controlled by oral drugs such as celebrex and IR codon, and injections such as tramadol and demerol. On the first postoperative day, the urinary catheter is removed and CPM (continuous passive motion) rehabilitation is started.
  Arms: Enhanced recovery after surgery (ERAS) patients

SUMMARY:
The purpose of this study is to analyze the effect of the ERAS(early recovery after surgery) protocol on total knee and hip arthroplasty compared to conventional standard protocol. Patients will be divided into two groups: ERAS protocol group and standard protocol group. On the day before the surgery, the patient group was randomly assigned by the researcher (research nurse) who did not participate in the surgical procedure. By comparing the clinical outcomes and quality of postoperative recovery of both groups, we could confirm the effect of ERAS protocol.

DETAILED DESCRIPTION:
The patients who underwent radiologic examination at Severance Hospital of Severance Hospital and who will received total knee arthroplasty or total hip arthroplasty due to primary degenerative osteoarthritis or osteonecrosis of femoral head. Patients will be divided into two groups: ERAS (early recovery after surgery) protocol group and standard protocol group. On the day before the surgery, the patient group was randomly assigned by the researcher (research nurse) who did not participate in the surgical procedure.

The patients in the ERAS group were given a pre-treatment drug [300 mg (gabapentin) and 10 mg oxycontin (oxycontin) and 2 mg prednisolone (prednisolone 10 mg)] on the evening before surgery. And pre-operative fasting should not exceed 6 hours, and clear liquid fasting should not exceed 2 hours. In addition, 400 ml of oral carbohydrate should be taken 2 to 4 hours before surgery to ensure adequate blood sugar and encourage regular diet (light meal) as soon as possible within a tolerable range after surgery. The initial pain after surgery is actively controlled by oral drugs such as celebrex and IR codon, and injections such as tramadol and demerol. On the first postoperative day, the urinary catheter is removed and CPM (continuous passive motion) rehabilitation is started.

On the other hand, in standard group, there is no medication as a pre-treatment drug. Patients should be fasted for 8 hours in both solid and liquid preoperatively. After the surgery, allow a small amount of clear liquid to remain at the 4-hour fasting period after the operation, and allow the fluid to start within a tolerable range after 4 hours. The urinary catheter is removed on the first postoperative day and CPM rehabilitation is started from the afternoon. Post-operative ambulation should begin as early as possible on the second postoperative day.

All patients will undergo anesthesia for general anesthesia or spinal anesthesia with a nerve block (adductor canal block or femoral nerve block). The quality of recovery index was assessed on the day before surgery and on the POD 1 quality of recovery score (QoR) 40 questionnaire. And the length of hospital stay, first eating time, first assisted walking time, and start of rehabilitation after surgery of all patients will be recorded. The number of times that need antiemetics due to nausea / vomiting during the hospitalization period will be recorded. After discharge from the hospital, the patient will visit outpatient clinic at 4 ± 2 weeks postoperatively and will be checked a physical examination such as the ROM of the knee. At 3 ± 1 months and 6 ± 1 months after surgery, VAS, WOMAC, AKS, knee ROM, and PF score of all patients would be checked in outpatients clinic. In addition, morbidity, complications, mortality, and re-admission before and up to 6 months after surgery would be recorded.

ELIGIBILITY:
Inclusion Criteria:

* 1. elective total knee arthroplasty for degenerative osteoarthritis
* 2. elective total hip arthroplasty for osteoarthritis of osteonecrosis of femoral head

Exclusion Criteria:

* 1. ASA class >3
* 2. severe medical comorbidities
* 3. inflammatory arthritis including rheumatoid arthritis
* 4. severe instability of knee or hip
* 5. revision surgery

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-05-10 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Quality of recovery score(QoR40) | 1 day before surgery
  Before surgery, QoR40 questionnaires will be used to compare the quality of recovery after anesthesia. QoR40 is a 40 items quality of recovery score that has been validated in a diverse group of patients. It is comprised of five dimensions which are physical comfort (12 items), emotional state (9 items), physical independence (5 items), psychological support (7 items), and pain (7 items). Each item of the questionnaire is graded on a five-point Likert scale, and the global QoR-40 scores range from 40 (extremely poor quality of recovery) to 200 (excellent quality of recovery).
Quality of recovery score(QoR40) | postoperative 1 day
  After surgery, QoR40 questionnaires will be used to compare the quality of recovery after anesthesia. QoR40 is a 40 items quality of recovery score that has been validated in a diverse group of patients. It is comprised of five dimensions which are physical comfort (12 items), emotional state (9 items), physical independence (5 items), psychological support (7 items), and pain (7 items). Each item of the questionnaire is graded on a five-point Likert scale, and the global QoR-40 scores range from 40 (extremely poor quality of recovery) to 200 (excellent quality of recovery).

SECONDARY OUTCOMES:
Length of hospital stay | From pre-surgery to discharge, up to 4 weeks
  The investigators will record the entire length of hospital stay.
First eating time | From pre-surgery to discharge, up to 4 weeks
  The investigators will record how soon the patients have started a normal meal, assisted walking and continuous passive movement rehabilitation after surgery.
First assisted walking time | From pre-surgery to discharge, up to 4 weeks
  The investigators will record how soon the patients have started a normal meal, assisted walking and continuous passive movement rehabilitation after surgery.
Start of rehabilitation(CPM) | From pre-surgery to discharge, up to 4 weeks
  The investigators will record how soon the patients have started a normal meal, assisted walking and continuous passive movement rehabilitation after surgery.
Mortality | up to 6 months after surgery
  The investigators will investigate mortality up to 6 months after surgery.
Morbidity | up to 6 months after surgery
  The investigators will investigate morbidity up to 6 months after surgery.
Postoperative surgical complication | up to 6 months after surgery
  The investigators will investigate postoperative complication of surgery up to 6 months after surgery.
Number of readmission | up to 6 months after surgery
  The investigators will investigate number of readmission up to 6 months after surgery.
Clinical score of total joint arthroplasty (VAS) | at postoperative 3±1 months
  The investigators will record the clinical score of total joint arthroplasty(VAS) at 3 months after surgery.
Clinical score of total joint arthroplasty (WOMAC) | at postoperative 3±1 months
  The investigators will record the clinical score of total joint arthroplasty(WOMAC, The Western Ontario and McMaster Universities Arthritis) at 3 months after surgery.
Clinical score of total joint arthroplasty (AKS) | at postoperative 3±1 months
  The investigators will record the clinical score of total joint arthroplasty(AKS, American knee society score) at 3 months after surgery.
Clinical score of total joint arthroplasty (knee ROM) | at postoperative 3±1 months
  The investigators will record the clinical score of total joint arthroplasty(knee ROM) at 3 months after surgery.
Clinical score of total joint arthroplasty (Patellofemoral score) | at postoperative 3±1 months
  The investigators will record the clinical score of total joint arthroplasty(Patellofemoral score) at 3 months after surgery.
Clinical score of total joint arthroplasty (Harris hip score) | at postoperative 3±1 months
  The investigators will record the clinical score of total joint arthroplasty(Harris hip score) at 3 months after surgery.
Clinical score of total joint arthroplasty (VAS) | at postoperative 6±1 months
  The investigators will record the clinical score of total joint arthroplasty(VAS) at 6 months after surgery.
Clinical score of total joint arthroplasty (WOMAC) | at postoperative 6±1 months
  The investigators will record the clinical score of total joint arthroplasty(WOMAC, The Western Ontario and McMaster Universities Arthritis) at 6 months after surgery.
Clinical score of total joint arthroplasty (AKS) | at postoperative 6±1 months
  The investigators will record the clinical score of total joint arthroplasty(AKS, American knee society score) at 6 months after surgery.
Clinical score of total joint arthroplasty (knee ROM) | at postoperative 6±1 months
  The investigators will record the clinical score of total joint arthroplasty(knee ROM) at 6 months after surgery.
Clinical score of total joint arthroplasty (Patellofemoral score) | at postoperative 6±1 months
  The investigators will record the clinical score of total joint arthroplasty(Patellofemoral score) at 6 months after surgery.
Clinical score of total joint arthroplasty (Harris hip score) | at postoperative 6±1 months
  The investigators will record the clinical score of total joint arthroplasty(Harris hip score) at 6 months after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Orthopedic Surgery, Yonsei University, College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No